CLINICAL TRIAL: NCT05123586
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Two-Arm, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of LY3361237 as a Treatment for Adults With At Least Moderately Active Systemic Lupus Erythematosus
Brief Title: A IMMA Master Protocol: A Study of LY3361237 in Participants With at Least Moderately Active Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18248; J1V-MC-BT01 (Other: Eli Lilly and Company); 2021-001406-30 (EudraCT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-11-17 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Autoimmune Disease; BTLA B and T Lymphocyte attenuator; Immune checkpoint; Inhibitory checkpoint agonist antibody; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3361237 (Experimental): Participants are administered LY3361237 subcutaneously (SC) and standard of care (SOC)
  Interventions: Drug: LY3361237
- Placebo (Placebo Comparator): Placebo administered SC and SOC given at matching intervals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3361237 — Administered SC
  Arms: LY3361237
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the efficacy and safety of LY3361237 in participants with at least moderately active systemic lupus erythematosus (SLE). Study will last up to 34 weeks and may include up to 15 visits.

ELIGIBILITY:
Inclusion Criteria:

* Are diagnosed with SLE at least 24 weeks before Day 1 of study
* Have documentation of having a score of 10 or more points on the European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) 2019 classification criteria for SLE
* Have a SLEDAI-2K score ≥6 at screening (Day 1) and clinical Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥4 (not including any items related to laboratory values) at randomization (Day 2)
* Must be receiving at least 1 background standard-of-care medication for SLE

Exclusion Criteria:

* Participants are excluded if they have received any of the following medications or therapies within the indicated timeframe prior to the randomization visit (Day 2).
* Are currently receiving oral corticosteroids at doses >20 mg per day of prednisone (or equivalent) or have adjusted the dosage of corticosteroids within 2 weeks before starting study treatment
* Have received parenteral corticosteroids within 12 weeks before starting study treatment or are expected to require parenteral corticosteroids during the study
* Have a current or recent acute, active infection
* Have had a serious, chronic, recurring conditions of herpes simplex, herpes zoster, recurring cellulitis, chronic osteomyelitis)
* Have human immunodeficiency virus (HIV) infection, hepatitis B virus (HBV), hepatitis C infection (HCV), active tuberculosis (TB)
* Have active fibromyalgia or active occurrence of an inflammatory condition that, in the investigator's opinion, would make it difficult to appropriately assess SLE activity for the purposes of this study
* Have experienced a cardiac event within 24 weeks to 12 months prior to screening
* Have a history of clinically significant or uncontrolled illness that in the opinion of the investigator could put the participant at risk to participate in the study
* Are, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide
* Are pregnant or are intending to become pregnant or to breastfeed at any time in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (50):
- United States (19):
  - Arizona Arthritis & Rheumatology Associates, P. C., Mesa, Arizona
  - Arizona Arthritis & Rheumatology Associates, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research - Sun City, Sun City, Arizona
  - Newport Huntington Med Grp, Huntington Beach, California
  - Desert Medical Advances, Rancho Mirage, California
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Ezy Medical Research, Miami, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Atlanta Research Center for Rheumatology, Marietta, Georgia
  - Qualmedica Research, LLC, Evansville, Indiana
  - Tekton Research, Inc, Wichita, Kansas
  - Clinvest Research LLC, Springfield, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina, Hillsborough, North Carolina
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Tekton Research, Inc., Moore, Oklahoma
  - Tekton Research, Inc, Austin, Texas
  - Rheumatology Center Of Houston, Houston, Texas
  - Houston Rheumatology & Arthritis Specialists, Katy, Texas
- Argentina (8):
  - Clínica Privada Independencia, Munro, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - APRILLUS Asistencia E Investigacion, CABA, Ciudad Autónoma de Buenos Aire
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Santa Fe Province
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - APRILLUS Asistencia E Investigacion, Ciudad Autónoma de Buenos Aire
  - DOM Centro de Reumatología, Ciudad Autónoma de Buenos Aire
  - CENUDIAB, Ciudad Autónoma de Buenos Aire
- Czechia (3):
  - Revmatologie.s.r.o., Brno, Brno-město
  - Artroscan, s.r.o., Ostrava, Moravskoslezský kraj
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (4):
  - Nouvel Hôpital Civil (NHC), Strasbourg, Alsace
  - Centre Hospitalier Regional D'Orleans, Orléans, Centre-Val de Loire
  - Centre Hospitalier Universitaire de Toulouse - Hôpital Purpan, Toulouse, Haute-Garo
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
- Mexico (4):
  - CIMAB SA de CV, Torreón, Coahuila
  - Centro Medico del Angel, Mexicali, Estado de Baja California
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara, Jalisco
  - Investigacion Biomedica para el Desarrollo de Fármacos S.A. de C.V., Zapopan, Jalisco
- Poland (4):
  - Twoja Przychodnia Poznanskie Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki Nr 2 im. dr J. Biziela w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - Nova Reuma Społka Partnerska, Bialystok, Podlaskie Voivodeship
- Puerto Rico (4):
  - Centro Reumatologico Caguas, Caguas, PR
  - GCM Medical Group, PSC - Hato Rey Site, San Juan, PR
  - Latin Clinical Trial Center, San Juan
  - Mindful Medical Research, San Juan
- Taiwan (4):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Tri-Service General Hospital, Taipei City, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan, Taoyuan
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
URL: http://vivli.org/

REFERENCES:
- See also: A IMMA Master Protocol: A Study of LY3361237 in Participants With at Least Moderately Active Systemic Lupus Erythematosus — https://trials.lillytrialguide.com/en-US/trial/3HWfOwLvzwF3K7DwjS0tkg

RESULTS

PARTICIPANT FLOW:
Groups:
- 450 Milligrams (mg) - LY3361237: Participants received 450 mg of LY3361237 administered subcutaneously (SC) every 2 weeks (Q2W) along with their usual Standard of Care (SOC) medication for 24 weeks.
- Placebo: Participants received placebo administered SC Q2W along with their usual SOC medication for 24 weeks.
Period: Overall Study
Arm/Group | 450 Milligrams (mg) - LY3361237 | Placebo
Started | 42 | 43
Received At Least 1 Dose of Study Drug | 42 | 43
Completed | 41 | 39
Not Completed | 1 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 450 mg - LY3361237: Participants received 450 mg of LY3361237 administered SC Q2W along with their usual SOC medication for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | 450 mg - LY3361237 | Placebo | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.1) | 43.3 (11.1) | 43.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 42 | 80
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 27 | 52
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 7 | 14
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 30 | 30 | 60
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 7 | 8 | 15
  United States | 18 | 19 | 37
  Taiwan | 3 | 2 | 5
  Poland | 6 | 7 | 13
  Mexico | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Arthritis and/or Rash at Baseline Who Achieve Remission of Arthritis and/or Rash
Description: Remission of arthritis and/or rash is defined by the following: if only arthritis is present at baseline, then the primary endpoint is met if arthritis is absent at Week 24; if only rash is present at baseline, then the primary endpoint is met if rash is absent at Week 24; if both arthritis and rash are present at baseline, then the primary endpoint is met if either arthritis, or rash, or both arthritis and rash are absent at Week 24.
Time Frame: Week 24
Population: All participants who received at least 1 dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 450 mg - LY3361237 | Placebo
Number analyzed (Participants) | 42 | 43
Percentage of participants | 11.9 | 20.9

2. Secondary Outcome: Percentage of Participants Who Achieve Systemic Lupus Erythematosus Disease Activity Index-4 (SLEDAI-4) Response
Description: Percentage of participants who achieved SLEDAI-4 response was assessed. A SLEDAI-4 response is defined as a ≥ 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score from baseline. The SLEDAI-2K score range is from a minimum of 0 to a maximum of 105 (higher scores represent higher disease activity).
Time Frame: Week 24
Population: All participants who received at least 1 dose of the study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 450 mg - LY3361237 | Placebo
Number analyzed (Participants) | 42 | 43
Percentage of participants | 9.5 | 16.3

3. Secondary Outcome: Percentage of Participants Who Achieve Systemic Lupus Erythematosus Responder Index-4 (SRI-4 Response)
Description: Percentage of participants who achieved SRI-4 response was assessed. SRI-4 measures reduction in SLE disease activity and is a composite measure that includes the SLE Disease Activity Index (SLEDAI-2K), British Isles Lupus Activity Group (BILAG) 2004 and Physician Global Assessment. It is defined as: 1) Reduction of ≥4 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in the Physician's Global Assessment of Disease Activity. The score range is from 0 to 100, with higher scores indicating greater disease activity.
Time Frame: Week 24
Population: All participants who received at least 1 dose of study drug and have evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 450 mg - LY3361237 | Placebo
Number analyzed (Participants) | 42 | 43
Percentage of participants | 9.5 | 16.3

4. Secondary Outcome: Pharmacokinetics (PK): Steady-state Trough Serum Concentration of LY3361237 at Week 24
Description: PK: Steady-state trough serum concentration of LY3361237 at Week 24 was assessed.
Time Frame: Week 24
Population: All participants who received at least one dose of LY3361237 and had evaluable PK data for this outcome.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | 450 mg - LY3361237
Number analyzed (Participants) | 21
micrograms per milliliter (μg/mL) | 144 (73.8)

ADVERSE EVENTS:
Time Frame: Baseline Up To 25 Weeks
Description: All participants who received at least 1 dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 450 mg - LY3361237 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 5/42 | 1/43
Other Adverse Events (participants affected / at risk) | 28/42 | 27/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 450 mg - LY3361237 (N=42) | Placebo (N=43)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 450 mg - LY3361237 (N=42) | Placebo (N=43)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polydactyly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 3 (3) | 0 (0)
Injection site bruising (General disorders) | 2 (6) | 0 (0)
Injection site erythema (General disorders) | 5 (14) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Injection site oedema (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 6 (97) | 3 (32)
Injection site reaction (General disorders) | 2 (21) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0/38 (0) | 1/42 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 4 (4) | 3 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Oral herpes (Infections and infestations) | 3 (3) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (5)
Urinary tract infection (Infections and infestations) | 4 (5) | 6 (6)
Vulvovaginal mycotic infection (Infections and infestations) | 0/38 (0) | 1/42 (1)
Vulvovaginitis (Infections and infestations) | 1/38 (1) | 0/42 (0)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Cardiolipin antibody positive (Investigations) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (9) | 1 (2)
Migraine (Nervous system disorders) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1/38 (1) | 0/42 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0/38 (0) | 1/42 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (4):
  • Study Protocol: Protocol ISA J1V-MC-BT01 (a) (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT05123586/Prot_000.pdf
  • Study Protocol: Master Protocol J1V-MC-IMMA (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT05123586/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan J1V-MC-BT01 Version 3 (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05123586/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan J1V-MC-IMMA Version 2 (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT05123586/SAP_003.pdf